CLINICAL TRIAL: NCT01736020
Title: Developing Anesthesia as PTSD Therapy
Brief Title: Developing Anesthesia as Post Traumatic Stress Disorder (PTSD) Therapy
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Southern California Institute for Research and Education (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); University of California, Irvine (Other)
Responsible Party: Principal Investigator, Michael Alkire, Associate Professor, Southern California Institute for Research and Education
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: MIRB 1007, UCI 2004-3707; R34MH087390 (NIH)
Record Dates: First submitted 2012-11-16; First posted 2012-11-29 (Estimated); Last update posted 2016-10-13 (Estimated); Status verified 2016-10

CONDITIONS: Healthy
MeSH Terms: interventions — Dexmedetomidine; Propofol; Ketamine; Nitrous Oxide

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Dexmedetomidine; Drug: Propofol; Drug: Ketamine; Drug: Nitrous Oxide; Drug: Placebo
- Dexmedetomidine (Experimental): Dexmedetomidine intravenous infusion during scan.
  Interventions: Drug: Dexmedetomidine
- Propofol (Experimental): Propofol intravenous infusion during scan.
  Interventions: Drug: Propofol
- Ketamine (Experimental): Ketamine intravenous infusion during scan.
  Interventions: Drug: Ketamine
- Nitrous Oxide (Experimental): Nitrous Oxide inhalation during scan.
  Interventions: Drug: Nitrous Oxide

INTERVENTIONS:
Drug: Dexmedetomidine — A low dose of dexmedetomidine is used during scanning after dose piloting outside the scanner for memory effects and tolerability.
  Arms: Dexmedetomidine; Placebo
Drug: Propofol — A low dose of propofol is used during scanning after dose piloting outside the scanner for memory effects and tolerability.
  Arms: Placebo; Propofol
Drug: Ketamine — A low dose of ketamine is used during scanning after dose piloting outside the scanner for memory effects and tolerability.
  Arms: Ketamine; Placebo
Drug: Nitrous Oxide — A low dose of nitrous oxide is used during scanning after dose piloting outside the scanner for memory effects and tolerability.
  Arms: Nitrous Oxide; Placebo
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This preclinical phase 1 development study in healthy volunteers seeks to identify if low doses of commonly used non-triggering anesthetic agents might have clinical utility for modulating emotional memory processing and to understand the nature of the brain mechanisms of drug action. Optimally, a drug, dose and brain mechanism of action will be identified that will form the foundation for future use in clinical studies of patients with PTSD.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults.
* Between the ages of 18 and 35.

Exclusion Criteria:

* Pregnancy.
* Left-handed.
* Unusual facial anatomy.
* History of esophageal reflux.
* Respiratory problems.
* Central nervous system disorders.
* Cardiovascular problems.
* Kidney disease.
* Diabetes.
* History of Substance abuse.
* History of adverse anesthetic reactions.
* Hepatitis.
* Failure to pass MRI screening questionnaire.
* Fear of small-enclosed spaces.
* Mental illness.
* Non-native English speakers.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 293 (Actual)
Dates: Start 2009-09; Primary Completion 2017-04 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
Number of events remembered | Day 4
  The proportion of items remembered in long-term memory 4 days after viewing emotional or neutral pictures.

SECONDARY OUTCOMES:
Event-related fMRI BOLD signals | Baseline
  Evoked fMRI responses to emotional and neutral pictures are measured and later correlated with subsequent memory performance.

OTHER OUTCOMES:
Tolerability | Baseline
  Subjective and objective measures of subject responses to the various agents are noted.

CONTACTS AND LOCATIONS:
Overall Officials: Michael T Alkire, MD, Principal Investigator — University of California, Irvine and Long Beach VA Medical Center
Locations (1):
- University of California, Irvine, Irvine, California, United States